CLINICAL TRIAL: NCT04920513
Title: Universal- Versus Guidelines-Directed Genetic Testing for Germline Pathogenic Variants Utilizing a Multi-Gene Panel for Inherited Cancers in Non-Western Society.
Status: Completed | Type: Observational
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Hikmat Abdel-Razeq, Professor, Chairman of department of medicine, Chief Medical officer, Deputy Director General, King Hussein Cancer Center
Other Study IDs: 21 KHCC 27
Record Dates: First submitted 2021-05-16; First posted 2021-06-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Genetic Predisposition
Keywords: Genetics
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators aim to study the pattern and frequency of pathogenic variants among ALL newly diagnosed cancer patients in a genetically distinct population.

Additionally, the investigators will study the uptake rate of "cascade family screening", frequency of pathogenic variants and barriers against testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age ≥ 18 years at time of cancer diagnosis
* Pathology proven diagnosis of cancer; any site, any stage (prior history of cancer is allowed)
* Jordanian nationality
* Willingness to participate
* Signed consent form

Exclusion Criteria:

* Major psychiatric disorder (defined as: patients followed by a psychiatrist and on antipsychotic medications)
* Non-Jordanian
* Patients with Leukemia, Lymphoma and Myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who fulfill the inclusion/exclusion criteria and are diagnosedat KHCC will be invited.
  A total of 3000 patients are estimated to participate
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of pathogenic or likely pathogenic germline variants among newly diagnosed cancer patients tested by universal multigene panel testing | 2021-2023
Number of participants with variants of uncertain significance (VUS) as assessed by universal multigene panel testing | 2021-2023
To determine the reasons/ Barriers for refusal of genetic cascade testing among newly diagnosed cancer patients. | 2021-2023

SECONDARY OUTCOMES:
Rate of cascade of family member testing of the participants with positive pathogenic mutation | 2021-2023
  The family of tested patients with pathogenic mutations will be offered the genetic testing
Prevalence of pathogenic or likely pathogenic mutations among tested family members of the participants with pathogenic mutations using the universal multigene panel | 2021-2023
Prevalence of variants of uncertain significance (VUS) among tested family members of participants with pathogenic mutations as assessed by universal multigene panel testing | 2021-2023
To determine the reasons/ Barriers for refusal of genetic cascade testing among family members of tested patients with pathogenic mutation | 2021-2023

CONTACTS AND LOCATIONS:
Overall Officials: Hikmat Abdel-Razeq, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Amman Governorate, Jordan